CLINICAL TRIAL: NCT01459562
Title: A Randomized Double-blinded Placebo Controlled Single Center Phase I Study of Escalating Single Intravenous Doses of NI-0501 in Healthy Volunteers
Brief Title: First in Human Study of an Anti-IFN Gamma Monoclonal Antibody in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Swedish Orphan Biovitrum (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Basic Science
Other Study IDs: NI-0501-03
Record Dates: First submitted 2011-10-17; First posted 2011-10-25 (Estimated); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Emapalumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- NI-0501 (Experimental)
  Interventions: Drug: NI-0501
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NI-0501
  Arms: NI-0501
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the safety, pharmacodynamic and pharmacokinetic profiles of a novel therapeutic drug when administered to healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* healthy adults between 18 and 50 years old
* non smokers
* able to adhere to study protocol requirements

Exclusion Criteria:

* any abnormal clinical safety laboratory parameters

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2011-09; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of escalating single IV doses of NI-0501. | AEs at: Study Day (SD) 1 pre-infusion, SD1 at 1, 2, 4, 8, 10, 12 hrs post infusion start, SD 2, SD 3, SD 5, SD 8, Wk 2, Wk 4, Wk 6, Wk 8

SECONDARY OUTCOMES:
Pharmacokinetics parameters, Determination of any pharmacodynamic effects, Immunogenicity of NI-0501 | PK/PD at: Study Day (SD) 1 pre-infusion, SD1 at 1, 2, 4, 8, 10 hrs post infusion start, SD 2, SD 3, SD 5, SD 8, Wk 2, Wk 4, Wk 6, Wk 8, Immunogenicity: SD1 pre-infusion, Wk 8

CONTACTS AND LOCATIONS:
Overall Officials: Steve Warrington, MD, Principal Investigator — HMR; Peter Dewland, MD, Principal Investigator — ICON plc
Locations (2):
- United Kingdom (2):
  - HMR, London
  - ICON, Manchester